CLINICAL TRIAL: NCT06152029
Title: Efficacy of a Temporary Peripheral Nerve Stimulation System in Patients With Osteoarthritis of the Knee
Brief Title: Temporary Peripheral Nerve Stimulation System for Osteoarthritis of the Knee
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left Advocate Health
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00104845; 23.135E (Other: Aurora IRB)
Record Dates: First submitted 2023-11-15; First posted 2023-11-30 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis
Keywords: Peripheral nerve stimulation; PNS
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with a temporary PNS system: These patients will receive a temporary PNS system for their knee pain secondary to osteoarthritis
  Interventions: Device: Temporary PNS system

INTERVENTIONS:
Device: Temporary PNS system — This system remains in place up to 60 days, then removed.
  Other Names: SPRINT PNS System

SUMMARY:
The purpose of this study is to demonstrate the treatment outcomes of patients with chronic knee pain secondary to osteoarthritis that have received a temporary peripheral nerve stimulation system.

ELIGIBILITY:
Inclusion Criteria:

* Age of 21 and older
* Will receive a temporary PNS system for the management of chronic knee pain secondary to osteoarthritis
* Be capable of subjective evaluation, able to read and understand English-written questionnaires, and able to read, understand and sign the written informed consent in English
* Be willing and capable of giving informed consent
* Be willing and able to comply with study-related requirements, procedures, and scheduled visits

Exclusion Criteria:

* No knee pain at rest
* Same nerve targeted for both Radiofrequency Ablation (RFA) and Peripheral Nerve Stimulation (PNS) in less than 6 months post RFA, if applicable
* Pregnancy
* History of repetitive skin infections
* Vulnerable populations (e.g., prisoners, minors, students, employees)
* Any other condition that may interfere with the ability to participate in a clinical trial (e.g., anatomy that may interfere with lead placement, nerve damage, compromised immune system, uncontrolled diabetes)
* Confounding conditions such as lumbar radiculopathy
* Deep brain stimulation system, implanted active cardiac implant (e.g. pacemaker of defibrillator), or any other implantable neuro-stimulator whose stimulus current pathway may overlap the SPRINT system.
* Be involved in an injury claim under current litigation
* Be a recipient of temporary Social Security Disability Insurance (SSDI) benefits due to chronic pain
* Have a pending or approved worker's compensation claim

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes patients with chronic knee pain secondary to osteoarthritis of the knee and will receive a temporary peripheral nerve stimulation device.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Average change from baseline to end of treatment in average pain intensity measured through BPI-SF item 5. | up to 60 days post lead placement

SECONDARY OUTCOMES:
Average change from baseline to end of treatment in health-related quality of life measured through PROMIS-29. | up to 60 days post lead placement
Average change from baseline to end of treatment in pain interference measured through BPI-SF. | up to 60 days post lead placement
Average change in chronic pain related medication intake at end of treatment compared to baseline in Morphine Miligram Equivalents (MME) | up to 60 days post lead placement
Overall patient global impression of change (PGIC) at end of treatment. | up to 60 days post lead placement
Overall incidence of lead migration/fracture at the end of treatment. | up to 60 days post lead placement
Average change from baseline to 7- and 30-days post-implant; and 6- and 12-months post-explant in average pain intensity measured through BPI-SF item 5. | 7 and 30 days post lead placement; and 6 and 12 month post lead pull
Average change from baseline to 6- and 12-months post-explant in health-related quality of life measured through PROMIS-29. | 7 and 30 days post lead placement; and 6 and 12 month post lead pull
Average change from baseline to 6- and 12-months post-explant in pain interference measured through BPI-SF. | 7 and 30 days post lead placement; and 6 and 12 month post lead pull
Overall patient global impression of change (PGIC) at 6 months and end of study. | 6 and 12 months post lead pull
Overall incidence of lead migration/fracture during the study. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Littlefield Lauren, MD, Principal Investigator — Aurora Medical Center Oshkosh - 855 N Westhaven Dr
Locations (2):
- United States (2):
  - Aurora Health Center, Fond du Lac, Wisconsin
  - Aurora Health Oshkosh, Oshkosh, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided